CLINICAL TRIAL: NCT06752538
Title: Assessment of Robotic Versus Laparoscopic Gastrectomy for Gastric Cancer Patients With Intraoperative Technical Complexity: A Multicenter Retrospective Study
Brief Title: Assessment of Robotic Versus Laparoscopic Gastrectomy for GC Patients With Intraoperative Technical Complexity
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: 2024KY216; 2024KY216 (Other: Fujian Medical University Union Hospital)
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Gastrectomy for Gastric Cancer; Robotic Surgical Procedures; Laparoscopic Surgical Procedures
Keywords: Surgical difficulty; Gastrectomy; Robotic; Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RG group: Patients undergoing robotic gastrectomy
- LG group: Patients undergoing laparoscopic gastrectomy

SUMMARY:
While robotic gastrectomy (RG) is increasingly used in gastric cancer surgery, its potential advantages over laparoscopic gastrectomy (LG) in Intraoperative technical complexity (ITC) cases remain debated.

DETAILED DESCRIPTION:
This retrospective cohort study included 3,534 patients with gastric cancer who underwent radical gastrectomy at eight high-volume hospitals. ITC was defined by any of the following criteria: operative time exceeding the third quartile, intraoperative estimated blood loss ≥ 400 mL, or conversion to open surgery. Propensity score matching (PSM) and inverse probability of treatment weighting (IPTW) were conducted to compare short- and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with postoperatively histologically confirmed T1-4aN0-3bM0 gastric adenocarcinoma who underwent RG or LG

Exclusion Criteria:

* Remnant gastric cancer
* Previous malignant
* ASA class >3
* Use of indocyanine green
* Neoadjuvant chemotherapy
* Loss to follow-up
* Combined resection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologically confirmed T1-4aN0-3bM0 gastric adenocarcinoma who underwent radical RG or LG between August 2016 and June 2019 at eight high-volume tertiary teaching hospitals in China
Sampling Method: Non-Probability Sample
Enrollment: 3534 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | Within 3 years after surgery
  Telephone follow-up

SECONDARY OUTCOMES:
recurrence | 36 months
  Telephone follow-up
Postoperative complications | 30 days after surgery
  Postoperative complications were evaluated according to the Clavien-Dindo classification and categorized as surgical or medical

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, PhD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No